CLINICAL TRIAL: NCT06931483
Title: The Efficacy and Safety of Transcranial Temporal Interference Stimulation (tTIS) Targeting the Right Globus Pallidus Internus (GPi) for Motor Symptoms in Patients With PD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yanghua Tian (Other)
Responsible Party: Sponsor-Investigator, Yanghua Tian, Vice President of Anhui Medical University, The Second Hospital of Anhui Medical University
Organization: The Second Hospital of Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AHMU-tTIS-PD
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Temporal Interference Stimulation; Parkinson's Disease; the Right Globus Pallidus Internus; Motor Symptoms
Keywords: temporal interference stimulation; Parkinson's Disease; motor symptoms; the right globus pallidus internus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real stimulation (Active Comparator): Participants will receive active tTIS for 10 days.
  Interventions: Device: Transcranial temporal interference stimulation (tTIS)
- sham stimulation (Sham Comparator): Participants will receive sham tTIS for 10 days.
  Interventions: Device: Sham transcranial temporal interference stimulation (tTIS)

INTERVENTIONS:
Device: Transcranial temporal interference stimulation (tTIS) — The total stimulation duration was 30 minutes, including a 30-second current ramp-up at the beginning and a 30-second ramp-down at the end.
  Arms: real stimulation
Device: Sham transcranial temporal interference stimulation (tTIS) — Sham stimulation had only 30 seconds of current ramping-up and ramping-down at the beginning and end of the stimulation, respectively, to simulate the sensation of actual stimulation.
  Arms: sham stimulation

SUMMARY:
To demonstrate that intervention targeting the right globus pallidus internus (GPi) using transcranial temporal interference stimulation can improve motor symptoms in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Each of patients received either 30-minute or sham tTIS of the right GPi. Before and immediately after the stimulation, participants completed the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS-III) in the "medication-on" state to assess the motor symptoms. MDS-UPDRS, HAMA and HAMD were assessed on intervention Day 1, Day 10 and 1-month follow-up and clinical efficacy was evaluated by comparing the scale scores before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the diagnostic criteria for Parkinson's disease in China (2016 version), diagnosed as PD by two neurologists;
2. Hoehn-Yahr stage 1.5-4;
3. Age > 50 years old;
4. No signs of moderate to severe depression: Beck Depression Inventory-II (BDI-II) score < 20;
5. No signs of dementia: Mini-Mental State Examination (MMSE) score > 21;
6. No change in medication regimen in the four weeks prior to enrollment;
7. Right-handed.

Exclusion Criteria:

1. History of other neuropsychiatric disorders;
2. History of alcohol or drug abuse;
3. Previous history of TMS or traditional TES treatment;
4. Presence of non-MRI compatible metal implants in the body, such as deep brain stimulation devices, pacemakers or stents.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | On intervention Day 1, Day 10 and 1-month follow-up.
  To assess the motor symptoms, participants completed the official Chinese version of MDS-UPDRS.The MDS-UPDRS-III includes 33 items, with scores ranging from 0 to 132. The subscores of MDS-UPDRS-III, including (1) rigidity (item 3.3), (2) bradykinesia (items 3.2, 3.4, 3.8, and 3.14), (3) tremor (items 3.15-3.18), and (4) axial signs (items 3.9-3.13), were also used as the secondary outcomes in the following analyses.

SECONDARY OUTCOMES:
emotional symptoms assessed by the HAMA | on intervention Day 1, Day 10 and 1-month follow-up
  The HAMA is a 14-item scale to measure the severity of anxiety symptoms, where each item is rated on a scale from 0 to 4. The HAMA total score ranges from 0 to 56, with lower scores indicating less anxiety symptoms.
emotional symptoms assessed by the HAMD | On intervention Day 1, Day 10 and 1-month follow-up.
  The HAMD is a clinic ian-administered depression assessment and consists of 17 items with a total score range from 0 to 54. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China